CLINICAL TRIAL: NCT02391077
Title: A Randomized, Open Label, Two Phase Trial, to Assess Various Antimicrobial Techniques for Reducing Bacterial Load Prior PrePex Removal
Brief Title: A Trial Assessing Efficacy of Various Antimicrobial Techniques for Reducing Bacterial Load
Acronym: RMC-11
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ministry of Health, Rwanda (Other Government)
Responsible Party: Principal Investigator, Vincent Mutabazi, Director of the Research Grants Unit, Ministry of Health, Rwanda
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RMC-11
Record Dates: First submitted 2015-02-15; First posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Disease Due to Gram-positive Bacteria
Keywords: PrePex; Male Circumcision; Bacterial Load
MeSH Terms: interventions — Povidone-Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Arm (No Intervention): Standard PrePex Procedure
- Arm 1 - Maximal intervention (Experimental): 1. Foreskin disinfection with Povidone-Iodine
  2. Application of 1gr of Antibiotic topical cream / ointment onto the exposed inner foreskin up to the coronal sulcus
  3. Daily washes with Chlorhexidine 1% (2-3 times a day), for 6 days
  Interventions: Other: Povidone-Iodine; Other: Antibiotic topical cream; Other: Chlorhexidine 1%
- Arm 2 - Medium intervention (Experimental): 1. Foreskin disinfection with Povidone-Iodine
  2. Application of 1gr of Antibiotic topical cream / ointment onto the exposed inner foreskin up to the coronal sulcus
  Interventions: Other: Povidone-Iodine; Other: Antibiotic topical cream

INTERVENTIONS:
Other: Povidone-Iodine — Foreskin disinfection with Povidone-Iodine
  Arms: Arm 1 - Maximal intervention; Arm 2 - Medium intervention
Other: Antibiotic topical cream — Application of 1gr of Antibiotic topical cream / ointment onto the exposed inner foreskin up to the coronal sulcus
  Arms: Arm 1 - Maximal intervention; Arm 2 - Medium intervention
Other: Chlorhexidine 1% — Daily washes with Chlorhexidine 1% (2-3 times a day), for 6 days
  Arms: Arm 1 - Maximal intervention

SUMMARY:
There is a potential of bacterial overgrowth under the foreskin in the sub-preputial space, therefore we would like to investigate possible techniques to reduce this potential.

DETAILED DESCRIPTION:
The PrePex device was accepted for the World Health Organization (WHO) list of prequalified male circumcision (MC) devices and was listed on 31 May 2013.

PrePex became the first medical device for adult male circumcision to receive WHO prequalification as an alternative to the conventional surgical circumcision methods already recognized by WHO.

Voluntary Medical Male Circumcision (VMMC) is a one-time, low cost intervention that shown to reduce men's risk of HIV infection by approximately 70 percent. The WHO recommends VMMC as part of a comprehensive package of HIV prevention services.

The PrePex compresses the foreskin causing ischemic necrosis. Due to the foreskin necrotic state, it is no longer possible for men to fully retract the skin and properly clean the sulcus and inner foreskin, the sub-preputial space normally has a low oxygen environment facilitating anaerobe growth, and following device placement the environment becomes more so leading to a higher bacterial load. This was suggested by reports of unpleasant odor following device placement and confirmed by laboratory test done by RHSP Uganda of swabs taken from inside the foreskin prior to device removal, results not yet published.

There is a potential of bacterial overgrowth under the foreskin in the sub-preputial space, therefore we would like to investigate possible techniques to reduce this potential.

This trial aims to validate the actions needed to minimize the probability of aerobic and anaerobic bacteria overgrowth once PrePex is introduced, and establish a safer procedure.

The trial encompasses different safe and known techniques, such as usage of anti-bacterial topical ointment, its objectives will be evaluated using laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Ages - 21 to 49 years
* Subject wants to be circumcised
* Uncircumcised
* Able to understand the study procedures and requirements
* Agrees to participate in either arm and to follow the hygiene and wound care instructions
* Agrees to have swab samples
* Agrees to abstain sexual intercourse for 6 weeks post device removal
* Agrees to abstain from masturbation for 2 weeks post device removal
* Agrees to return to the health care facility for follow-up visits (or as instructed) after his circumcision
* Subject able to comprehend and freely give informed consent for participation in this study and is considered by the investigator to have good compliance for the study
* Subject agrees to anonymous video and photographs of the procedure and follow up visits.

Exclusion Criteria:

* Active genital infection, anatomic abnormality or other condition, which in the opinion of the investigator prevents the subject from undergoing a circumcision
* Subject with the following diseases/conditions: phimosis, paraphimosis, warts under the prepuce, torn or tight frenulum, narrow prepuce, hypospadias, epispadias
* Known bleeding / coagulation abnormality, uncontrolled diabetes, by questionnaire
* Known allergy to Betadin-Iodine
* Known allergy to antibiotics containing Bacitracin, Neomycin and Polymixin
* Subject who have an abnormal penile anatomy or any penile diseases
* Subject that to the opinion of the investigator is not a good candidate
* Subject does not agree to anonymous video and photographs of the procedure and follow up visits.

Ages: 21 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
The semi quantitative count of bacteria on days 0 and 7 | Days 0 and 7

SECONDARY OUTCOMES:
Placement preparation technique as a measure of reduction of preputial space bacterial load | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Mutabazi, M.D., Principal Investigator — Ministry of Health, Rwanda
Locations (1):
- Kanombe Military Hospital, Kigali, Kigali, Rwanda

REFERENCES:
- See also: Rwanda Biomedical Centre — http://www.rbc.gov.rw/